CLINICAL TRIAL: NCT01678937
Title: Immune Tolerance and Alloreactivity in Liver Transplant Recipients on Different Monotherapy Immunosuppressive Agents
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Northwestern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Josh Levitsky, Associate Professor in Medicine-Hepatology, Northwestern University
Other Study IDs: 1783-011
Record Dates: First submitted 2011-07-08; First posted 2012-09-05 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Liver Transplant Rejection; Immunosuppression
Keywords: Immunosuppression
MeSH Terms: interventions — Sirolimus; Cyclosporine; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood tests: Monotherapy patients
  1. Regulatory/Suppressor Cells (CD4+CD25+FOXP3+CD127low; and CD8+ CD28-FOXP3+CD127low cells).
  2. Dendritic cell assays: myeloid vs. lymphoid (CD11c; CD123); maturation and ability to process antigens (CD83; CD205); markers that have been shown to induce regulatory T cells (ILT3; ILT4).
  3. Soluble HLA G
  Blood tests: Conversion patients
  1. Regulatory/Suppressor Cells (CD4+CD25+FOXP3+CD127low; and CD8+ CD28-FOXP3+CD127low cells).
  2. Dendritic cell assays: myeloid vs. lymphoid (CD11c; CD123); maturation and ability to process antigens (CD83; CD205); markers that have been shown to induce regulatory T cells (ILT3; ILT4),
  3. Soluble HLA G, and
  4. Liver function and drug levels.
  Blood tests: Healthy controls (same tests as Monotherapy Group)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control Group: Ten Healthy individuals will have blood drawn (4 green top tubes(40 ml = 8 tsp.)) at one time point at Northwestern for control purposes. Blood will be drawn to conduct the following tests:
  1. Dendritic cell assays: myeloid vs. lymphoid (CD11c; CD123); maturation and ability to process antigens (CD83; CD205); markers that have been shown to induce regulatory T cells (ILT3; ILT4).
  2. Regulatory/Suppressor Cells (CD4+CD25+FOXP3+CD127low; and CD8+ CD28- FOXP3+CD127low cells), and
  3. HLA microchimerism & HLA G.
  Interventions: Procedure: Blood Draw from Control Subjects
- Monotherapy Group: Monotherapy patients [cyclosporine (CyA) (10 patients), Tacrolimus (5 patients), mycophenolate mofetil (MMF) (10 patients), rapamycin (10 patients)]: Blood will be drawn at one time point (4 green top tubes (40 ml = 8 tsp.)) to conduct the following tests:
  1. Dendritic cell assays: myeloid vs. lymphoid (CD11c; CD123); maturation and ability to process antigens (CD83; CD205); markers that have been shown to induce regulatory T cells (ILT3; ILT4).
  2. Regulatory/Suppressor Cells (CD4+CD25+FOXP3+CD127low; and CD8+ CD28- FOXP3+CD127low cells), and
  3. HLA microchimerism & HLA G.
  Interventions: Procedure: Blood Draw - CyA; Procedure: Blood Draw - Tacrolimus; Procedure: Blood Draw - MMF; Procedure: Blood Draw - Rapamycin
- Conversion Group: Ten CNI monotherapy/dual therapy (CNI + MMF) patients pre-selected for conversion to rapamycin or wean to MMF monotherapy. Assays performed 2 weeks prior to conversion, 3-6 months following successful conversion. Liver function/drug levels monitored weekly during conversion until stable levels achieved. Patients converting from CNI monotherapy to rapamycin monotherapy (2-4 wks.): CNI discontinued when 2 therapeutic rapamycin levels (5-10) reached, graft function stable (clinical care protocol). MMF conversion: MMF dose slowly increased to 3 g/day (max.) while CNI therapy reduced by 1-2 mg/day (FK506) or 25-50 mg/day (CyA) monthly until CNI discontinued (1-6 months) (clinical care protocol). Monthly liver function/drug levels performed after successful conversion (standard of care).
  Interventions: Procedure: Blood Draw - Rapamycin

INTERVENTIONS:
Procedure: Blood Draw - Rapamycin — Ten calcineurin-inhibitors (CNI) monotherapy or dual therapy (CNI+MMF) patients will have blood taken (40 ml=8 tsp.) 2 wks. prior to conversion, 3-6 months post successful conversion. 1) Regulatory/Suppressor Cells (CD4+CD25+FOXP3+CD127low; and CD8+ CD28-FOXP3+CD127low cells). 2) Dendritic cell assays: myeloid vs. lymphoid (CD11c; CD123); maturation and ability to process antigens (CD83; CD205); markers shown to induce regulatory T cells (ILT3; ILT4), 3) Soluble HLA G, and 4) Liver function/drug levels. If problems develop during conversion (e.g. acute rejection, significant drug side effects) requiring discontinuation of rapamycin, MMF and/or reversion to CNI therapy, assays will not be performed. Monthly liver function/drug levels performed after successful conversion (standard of care).
  Other Names: Sirolimus
  Groups: Conversion Group
Procedure: Blood Draw from Control Subjects — Ten healthy individuals will have blood drawn (40 ml = 8 teaspoons (tsps.)).Blood will be drawn at one time point for the following:
  * Dendritic cell assays: myeloid vs. lymphoid (CD11c; CD123); maturation and ability to process antigens (CD83; CD205); markers that have been shown to induce regulatory T cells (ILT3; ILT4).
  * Regulatory/Suppressor Cells (CD4+CD25+FOXP3+CD127low; and CD8+ CD28- FOXP3+CD127low cells).
  * HLA microchimerism & HLA G
  Groups: Control Group
Procedure: Blood Draw - CyA — Blood drawn from 10 patients on cyclosporine (CyA) (40 ml = 8 tsp.)). Blood will be drawn at one time point for the following:
  * Dendritic cell assays: myeloid vs. lymphoid (CD11c; CD123); maturation and ability to process antigens (CD83; CD205); markers that have been shown to induce regulatory T cells (ILT3; ILT4).
  * Regulatory/Suppressor Cells (CD4+CD25+FOXP3+CD127low; and CD8+ CD28- FOXP3+CD127low cells).
  * HLA microchimerism & HLA G
  Other Names: cyclosporine
  Groups: Monotherapy Group
Procedure: Blood Draw - Tacrolimus — Blood drawn from 5 patients on Tacrolimus (40 ml = 8 tsp.) at one time point for the following:
  * Dendritic cell assays: myeloid vs. lymphoid (CD11c; CD123); maturation and ability to process antigens (CD83; CD205); markers that have been shown to induce regulatory T cells (ILT3; ILT4).
  * Regulatory/Suppressor Cells (CD4+CD25+FOXP3+CD127low; and CD8+ CD28- FOXP3+CD127low cells).
  * HLA microchimerism & HLA G
  Other Names: Tacrolimus
  Groups: Monotherapy Group
Procedure: Blood Draw - MMF — Blood will be drawn from 10 patients on mycophenolate mofetil (MMF) (40 ml or the equivalent of 8 teaspoons). Blood will be drawn at one time point for the following analysis:
  * Dendritic cell assays: myeloid vs. lymphoid (CD11c; CD123); maturation and ability to process antigens (CD83; CD205); markers that have been shown to induce regulatory T cells (ILT3; ILT4).
  * Regulatory/Suppressor Cells (CD4+CD25+FOXP3+CD127low; and CD8+ CD28- FOXP3+CD127low cells).
  * HLA microchimerism & HLA G
  Other Names: mycophenolate mofetil
  Groups: Monotherapy Group
Procedure: Blood Draw - Rapamycin — Blood drawn from 10 patients on rapamycin (40 ml = 8 tsp.)) at one time point for the following:
  * Dendritic cell assays: myeloid vs. lymphoid (CD11c; CD123); maturation and ability to process antigens (CD83; CD205); markers that have been shown to induce regulatory T cells (ILT3; ILT4).
  * Regulatory/Suppressor Cells (CD4+CD25+FOXP3+CD127low; and CD8+ CD28- FOXP3+CD127low cells).
  * HLA microchimerism & HLA G
  Other Names: Rapamycin
  Groups: Monotherapy Group

SUMMARY:
This study is being done with the purpose of trying to understand if and why transplant recipients may develop tolerance to their transplanted organ. Tolerance means being able to lower or take away immunosuppression (anti-rejection medications) without causing organ rejection.

DETAILED DESCRIPTION:
Life-long immunosuppressive therapy is typically required in the majority of liver allograft recipients. In the early years of liver transplantation (LT), the majority of deaths occurred secondary to graft loss from acute or chronic rejection despite immunosuppression (IS). With the advent of more powerful and specific IS agents, e.g. calcineurin-inhibitors (CNIs) cyclosporine (CyA) and tacrolimus (TAC), graft rejection rates significantly declined and short and long term graft/patient survival dramatically improved. However, along with the advance in survival rates came the adverse effects of long term immunosuppression (IS), e.g. morbidity and mortality from cardiovascular events, renal insufficiency, infectious complications, recurrent viral hepatitis and malignancy. These events are exacerbated by pre-existing conditions and an aging transplant population. Immunosuppression tapering or withdrawal could lower the incidence of these complications and improve long term graft and patient survival.

Therefore, the study proposed is a laboratory investigation (using blood samples collected from the subjects) comparing immune tolerance and alloreactivity profiles in LT recipients on monotherapy IS or converted to rapamycin monotherapy, to determine tolerogenic properties of the different IS agents. Knowledge of these properties would support the need for specific IS therapy to promote immune tolerance and consider IS withdrawal.

Monotherapy patients will be identified by the organ transplant database and medical charts at Northwestern. Patients will be invited to participate in the study and asked to undergo venipunctures for our analysis. Patient demographics, laboratories and other clinical data will be recorded. Patients on CNI monotherapy are continuously being identified for conversion to rapamycin monotherapy during clinic visits or chart reviews at Northwestern. Patients are selected for conversion due to significant CNI side effects, e.g. chronic kidney disease (creatinine clearance < 50 in the absence of significant proteinuria > 1g, poorly controlled diabetes mellitus/hypertension/hyperlipidemia, peripheral neuropathy). In general, patients are converted from CNIs to rapamycin over 2-3 weeks once therapeutic rapamycin levels are achieved.

Study procedures will be carried out by the investigators and associated personnel. Patients will be assigned a number in numerical order, to remove patient identifiers from the data analysis. A separate screening/enrollment log will be kept separate from the data. Baseline characteristics of the patients will be recorded: age, sex, liver disease, past medical history, history of acute rejection or other graft dysfunction, other post-LT complications, previous and current IS regimens. Monotherapy patients (10 from CyA, Tacrolimus, and MMF; 5 rapamycin) will be identified as above and asked to participate. Blood will be drawn at one time point for the following analysis:

* Dendritic cell assays: myeloid vs. lymphoid (CD11c; CD123); maturation and ability to process antigens (CD83; CD205); markers that have been shown to induce regulatory T cells (ILT3; ILT4).
* Regulatory/Suppressor Cells (CD4+CD25+FOXP3+CD127low; and CD8+ CD28- FOXP3+CD127low cells).
* HLA microchimerism & HLA G

Ten patients who have been pre-selected for rapamycin conversion will have the above assays performed two weeks prior to conversion and 3-6 months following conversion. They will also have liver function and drug level tests.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Orthotopic or Living-Related liver transplant (LT) recipient
* Monotherapy patients: > 6 months with stable graft function on current monotherapy (CNI, MMF, or rapamycin)
* Converting patients: CNI therapy converting to rapamycin or MMF monotherapy and > 6 months of stable graft function.
* >1 years post-LT without an acute rejection episode or chronic rejection
* Normal liver function tests (no recurrent HCV, chronic rejection, autoimmune hepatitis, etc.)
* No history of induction or lymphocyte depletion therapy

Exclusion Criteria:

* Multi-visceral organ recipients
* Graft dysfunction of any etiology
* Inadequate follow-up or available outcomes
* Unable to understand, sign or ask questions regarding the informed consent process and protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Liver transplant patients converting on stable IS monotherapy or undergoing conversion to rapamycin or MMF monotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2007-09; Primary Completion 2008-05 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Track interval outcome measures for development of higher percentages of FOXP3+ T1 regulatory cells in stable liver transplant recipients on rapamycin or MMF monotherapy compared to CNI monotherapy. | Two weeks prior to conversion, Months 3 & 6 following conversion
  * Dendritic cell assays: myeloid vs. lymphoid (CD11c; CD123); maturation and ability to process antigens (CD83; CD205); markers that have been shown to induce regulatory T cells (ILT3; ILT4).
  * Regulatory/Suppressor Cells (CD4+CD25+FOXP3+CD127low; and CD8+ CD28- FOXP3+CD127low cells).
  * Liver function and drug levels.
Track interval outcome measures for development of higher percentages of FOXP3+ T regulatory cells in liver transplant recipients after conversion from CNI to rapamycin comparing to MMF monotherapy. | Two weeks prior to conversion, Months 3 & 6 following conversion
  * Dendritic cell assays: myeloid vs. lymphoid (CD11c; CD123); maturation and ability to process antigens (CD83; CD205); markers that have been shown to induce regulatory T cells (ILT3; ILT4).
  * Regulatory/Suppressor Cells (CD4+CD25+FOXP3+CD127low; and CD8+ CD28- FOXP3+CD127low cells).

SECONDARY OUTCOMES:
Track interval outcome measures for development of higher percentages of immunophenotypic markers associated with regulatory T cell production in stable liver transplant recipients on rapamycin or MMF monotherapy compared to CNI monotherapy. | Two weeks prior to conversion, Months 3 & 6 following conversion
  * Dendritic cell assays: myeloid vs. lymphoid (CD11c; CD123); maturation and ability to process antigens (CD83; CD205); markers that have been shown to induce regulatory T cells (ILT3; ILT4).
  * Regulatory/Suppressor Cells (CD4+CD25+FOXP3+CD127low; and CD8+ CD28- FOXP3+CD127low cells).
  * HLA microchimerism & HLA G (dendritic cell ratios, soluble HLA G)
  * Liver function and drug levels.
Track interval outcome measures for development of higher percentages of immunophenotypic markers associated with regulatory T cell production in liver transplant recipients after conversion from CNI to rapamycin or MMF monotherapy. | Two weeks prior to conversion, Months 3 & 6 following conversion
  * Dendritic cell assays: myeloid vs. lymphoid (CD11c; CD123); maturation and ability to process antigens (CD83; CD205); markers that have been shown to induce regulatory T cells (ILT3; ILT4).
  * Regulatory/Suppressor Cells (CD4+CD25+FOXP3+CD127low; and CD8+ CD28- FOXP3+CD127low cells).
  * HLA microchimerism & HLA G (dendritic cell ratios, soluble HLA G)(hypertension, hyperlipidemia, renal insufficiency, diabetes, neuropathy)
Document improvement in adverse CNI side effects after conversion to rapamycin or MMF monotherapy, comparing designated time points. | Two weeks prior to conversion, Months 3 & 6 following conversion
  CNI side effects - hypertension, hyperlipidemia, renal insufficiency, diabetes, neuropathy. Review liver function and drug levels at designated time points.
Document the development of any adverse rapamycin or MMF side effects after conversion, comparing designated time points. | Two weeks prior to conversion, Months 3 & 6 following conversion
  Document Rapamycin side effects - oral ulcers, edema, pancytopenia, gastrointestinal dysfunction; or MMF side effects - pancytopenia, gastrointestinal dysfunction. Review liver function and drug levels at designated time points.

CONTACTS AND LOCATIONS:
Overall Officials: Josh Levitsky, MD, Principal Investigator — Northwestern University, Northwestern Memorial Hospital, Northwestern Medical Faculty Foundation
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Sayegh MH, Carpenter CB. Transplantation 50 years later--progress, challenges, and promises. N Engl J Med. 2004 Dec 23;351(26):2761-6. doi: 10.1056/NEJMon043418. No abstract available. PMID 15616214
- [Background] Takatsuki M, Uemoto S, Inomata Y, Egawa H, Kiuchi T, Fujita S, Hayashi M, Kanematsu T, Tanaka K. Weaning of immunosuppression in living donor liver transplant recipients. Transplantation. 2001 Aug 15;72(3):449-54. doi: 10.1097/00007890-200108150-00016. PMID 11502975
- [Background] Tisone G, Orlando G, Cardillo A, Palmieri G, Manzia TM, Baiocchi L, Lionetti R, Anselmo A, Toti L, Angelico M. Complete weaning off immunosuppression in HCV liver transplant recipients is feasible and favourably impacts on the progression of disease recurrence. J Hepatol. 2006 Apr;44(4):702-9. doi: 10.1016/j.jhep.2005.11.047. Epub 2006 Jan 4. PMID 16473433
- [Background] Girlanda R, Rela M, Williams R, O'Grady JG, Heaton ND. Long-term outcome of immunosuppression withdrawal after liver transplantation. Transplant Proc. 2005 May;37(4):1708-9. doi: 10.1016/j.transproceed.2005.03.070. PMID 15919439
- [Background] Hurwitz M, Desai DM, Cox KL, Berquist WE, Esquivel CO, Millan MT. Complete immunosuppressive withdrawal as a uniform approach to post-transplant lymphoproliferative disease in pediatric liver transplantation. Pediatr Transplant. 2004 Jun;8(3):267-72. doi: 10.1111/j.1399-3046.2004.00129.x. PMID 15176965
- [Background] Oike F, Yokoi A, Nishimura E, Ogura Y, Fujimoto Y, Kasahara M, Kaihara S, Kiuchi T, Egawa H, Uemoto S, Tanaka K. Complete withdrawal of immunosuppression in living donor liver transplantation. Transplant Proc. 2002 Aug;34(5):1521. doi: 10.1016/s0041-1345(02)02980-9. No abstract available. PMID 12176465
- [Background] Lerut J, Sanchez-Fueyo A. An appraisal of tolerance in liver transplantation. Am J Transplant. 2006 Aug;6(8):1774-80. doi: 10.1111/j.1600-6143.2006.01396.x. PMID 16889539
- [Background] Mazariegos GV, Reyes J, Marino I, Flynn B, Fung JJ, Starzl TE. Risks and benefits of weaning immunosuppression in liver transplant recipients: long-term follow-up. Transplant Proc. 1997 Feb-Mar;29(1-2):1174-7. doi: 10.1016/s0041-1345(96)00535-0. No abstract available. PMID 9123261
- [Background] Mazariegos GV, Reyes J, Marino IR, Demetris AJ, Flynn B, Irish W, McMichael J, Fung JJ, Starzl TE. Weaning of immunosuppression in liver transplant recipients. Transplantation. 1997 Jan 27;63(2):243-9. doi: 10.1097/00007890-199701270-00012. PMID 9020325
- [Background] Donckier V, Troisi R, Le Moine A, Toungouz M, Ricciardi S, Colle I, Van Vlierberghe H, Craciun L, Libin M, Praet M, Noens L, Stordeur P, Andrien M, Lambermont M, Gelin M, Bourgeois N, Adler M, de Hemptinne B, Goldman M. Early immunosuppression withdrawal after living donor liver transplantation and donor stem cell infusion. Liver Transpl. 2006 Oct;12(10):1523-8. doi: 10.1002/lt.20872. PMID 17004249
- [Background] Mazariegos GV, Zahorchak AF, Reyes J, Ostrowski L, Flynn B, Zeevi A, Thomson AW. Dendritic cell subset ratio in peripheral blood correlates with successful withdrawal of immunosuppression in liver transplant patients. Am J Transplant. 2003 Jun;3(6):689-96. doi: 10.1034/j.1600-6143.2003.00109.x. PMID 12780560
- [Background] Wong T, Nouri-Aria KT, Devlin J, Portmann B, Williams R. Tolerance and latent cellular rejection in long-term liver transplant recipients. Hepatology. 1998 Aug;28(2):443-9. doi: 10.1002/hep.510280223. PMID 9696010
- [Background] Devlin J, Doherty D, Thomson L, Wong T, Donaldson P, Portmann B, Williams R. Defining the outcome of immunosuppression withdrawal after liver transplantation. Hepatology. 1998 Apr;27(4):926-33. doi: 10.1002/hep.510270406. PMID 9537430
- [Background] Woltman AM, de Fijter JW, Kamerling SW, Paul LC, Daha MR, van Kooten C. The effect of calcineurin inhibitors and corticosteroids on the differentiation of human dendritic cells. Eur J Immunol. 2000 Jul;30(7):1807-12. doi: 10.1002/1521-4141(200007)30:73.0.CO;2-N. PMID 10940869
- [Background] Koenen HJ, Fasse E, Joosten I. Cyclosporine preserves the anergic state of human T cells induced by costimulation blockade in vitro. Transplantation. 2005 Aug 27;80(4):522-9. doi: 10.1097/01.tp.0000172217.97072.54. PMID 16123728
- [Background] Szabo G, Gavala C, Mandrekar P. Tacrolimus and cyclosporine A inhibit allostimulatory capacity and cytokine production of human myeloid dendritic cells. J Investig Med. 2001 Sep;49(5):442-9. doi: 10.2310/6650.2001.33789. PMID 11523700
- [Background] Battaglia M, Stabilini A, Roncarolo MG. Rapamycin selectively expands CD4+CD25+FoxP3+ regulatory T cells. Blood. 2005 Jun 15;105(12):4743-8. doi: 10.1182/blood-2004-10-3932. Epub 2005 Mar 3. PMID 15746082
- [Background] Battaglia M, Stabilini A, Draghici E, Gregori S, Mocchetti C, Bonifacio E, Roncarolo MG. Rapamycin and interleukin-10 treatment induces T regulatory type 1 cells that mediate antigen-specific transplantation tolerance. Diabetes. 2006 Jan;55(1):40-9. PMID 16380475
- [Background] Mehling A, Grabbe S, Voskort M, Schwarz T, Luger TA, Beissert S. Mycophenolate mofetil impairs the maturation and function of murine dendritic cells. J Immunol. 2000 Sep 1;165(5):2374-81. doi: 10.4049/jimmunol.165.5.2374. PMID 10946260
- [Background] Gregori S, Casorati M, Amuchastegui S, Smiroldo S, Davalli AM, Adorini L. Regulatory T cells induced by 1 alpha,25-dihydroxyvitamin D3 and mycophenolate mofetil treatment mediate transplantation tolerance. J Immunol. 2001 Aug 15;167(4):1945-53. doi: 10.4049/jimmunol.167.4.1945. PMID 11489974
- [Background] Nikolaeva N, Bemelman FJ, Yong SL, van Lier RA, ten Berge IJ. Rapamycin does not induce anergy but inhibits expansion and differentiation of alloreactive human T cells. Transplantation. 2006 Feb 15;81(3):445-54. doi: 10.1097/01.tp.0000194860.21533.b9. PMID 16477233
- See also: PMID: 19141306 — http://www.ncbi.nlm.nih.gov/pubmed